CLINICAL TRIAL: NCT05642481
Title: Therapeutic Drug Monitoring to oPtimize ANtiretroviral regimeNs in HIV-infected Women Who wAnt to Breastfeed
Acronym: PANNA-B TDM
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Amsterdam University Medical Center (Other); Erasmus Medical Center (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: PANNA-B TDM
Record Dates: First submitted 2022-11-09; First posted 2022-12-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-04

CONDITIONS: HIV-1-infection
Keywords: Breastfeeding; Therapeutic drug monitoring; Breast milk to maternal plasma ratio; Antiretroviral therapy
MeSH Terms: conditions — Breast Feeding | interventions — Drug Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — breastmilk, maternal plasma and infant plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antiretroviral drugs with marketing authorisation in Europe: This study includes subjects who already take antiretroviral drugs to treat HIV-1 with a marketing authorisation in Europe. These drugs already have a marketing authorisation and are prescribed by the treating physician of the subject. No adjustments to their treating regimen are made in order to participate in this study. All antiretrovirals with a marketing authorisation in Europe are eligible for inclusion in this study, but most subjects are expected to use a backbone of nucleoside reverse transcriptase inhibitors combined with either dolutegravir, raltegravir, darunavir or rilpivirine
  Interventions: Diagnostic Test: Therapeutic drug monitoring in plasma of mother and child and in breastmilk

INTERVENTIONS:
Diagnostic Test: Therapeutic drug monitoring in plasma of mother and child and in breastmilk — Measurement of drug concentration in plasma of mother and if possible of child and in breastmilk

SUMMARY:
This is a prospective, multi-center, longitudinal, mother-infant pair, therapeutic drug monitoring study. The aim of this study is to determine concentrations of antiretroviral drugs in plasma and breastmilk in people living with HIV who chose to breastfeed while using antiretrovirals. At a planned hospital visit an extra maternal blood sample (1 to 2 per visit) and extra infant blood sample (1 per visit) will be collected, as well as a breastmilk sample (1 to 2 per visit). Ideally, sample collection will take place at least during the 1, 3 and 6 month post partum follow up visit. Measured concentrations will be used to calculate milk to plasma ratios, relative and absolute infant dosages.

ELIGIBILITY:
Inclusion criteria

* Patients of at least 18 years of age at the moment of screening
* Patients with HIV-1 as documented with positive HIV antibody test, HIV RNA of antigen test
* Patients breastfeeding their infant
* Patients using antiretrovirals for the treatment of HIV-1 with a marketing authorisation in Europe (table 1 in Appendix)
* Patients using current antiretrovirals for a minimum of 2 weeks to assure drug concentrations are in steady state
* Patients who are able and willing to sign an informed consent

Exclusion Criteria:

No exclusion criteria will be used at the screening for the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women living with HIV using antiretroviral medication who chose to breastfeed their child
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Breastmilk to maternal plasma ratio | 6 months post partum
  Total concentration of antiretrovirals in breastmilk and plasma of the mother at a single time point to determine milk to plasma ratio.

SECONDARY OUTCOMES:
Absolute infant dose | 6 months post partum
  (AID; µg/kg/day) = Cmilk * Vmilk
Relative infant dose | 6 months post partum
  Dosage infant (AID)/dosage mother
Comparison of absolute infant dose to approved pediatric dose | 6 months post partum
  For agents approved for pediatric use the absolute infant dose is compared to the approved pediatric dose (abacavir, emtricitabine, lamivudine, zidovudine, efavirenz, nevirapine, atazanavir, lopinavir, maraviroc, dolutegravir, raltegravir, ritonavir)
Viral load in breastmilk | 6 months post partum
  HIV RNA (copies/ml)

OTHER OUTCOMES:
Adverse events in infant | At every follow up visit (1,2,3,4,5,6 months post partum)
  As reported by the parents/caregivers and/or paediatrician
The place of the infant in population-specific percentile distributions of weight for age | At every follow up visit (1,2,3,4,5,6 months post partum)
HIV RNA in infant | At every follow up visit (1,2,3,4,5,6 months post partum)
  (copies/ml)
Adverse events in mother | At every follow up visit (1,2,3,4,5,6 months post partum)
  As reported by mother and/or treating physician
Kidney function | At every follow up visit (1,2,3,4,5,6 months post partum)
  (estimated glomerular filtration rate - KDIGO)
Alanine aminotranferase in mother | At every follow up visit (1,2,3,4,5,6 months post partum)
Bilirubin in mother | At every follow up visit (1,2,3,4,5,6 months post partum)
Hemoglobin in mother | At every follow up visit (1,2,3,4,5,6 months post partum)
HIV RNA in mother | At every follow up visit (1,2,3,4,5,6 months post partum)
  copies/ml

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - Amsterdamumc, Amsterdam, North Holland
  - Erasmusmc, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided